CLINICAL TRIAL: NCT01583491
Title: Evaluation of Platelet Rich Fibrin Efficacy on Reduction of Periodontal Problems
Brief Title: Evaluation of Platelet Rich Fibrin on Reduction of Periodontal Problems After Surgical Removal of Mandibular Third Molar
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Majid Eshghpour (Other)
Responsible Party: Sponsor-Investigator, Majid Eshghpour, assistant professor, Mashhad University of Medical Sciences
Organization: Mashhad University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 900093
Record Dates: First submitted 2011-12-07; First posted 2012-04-24 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Mastication Disorder
Keywords: platelet rich fibrin; mandibular third molar; periodontal problem
MeSH Terms: interventions — Prolactin-Releasing Hormone; Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prf group.peridontal problem (Active Comparator): prf insert into surgical site immediate after surgery
  Interventions: Procedure: autologous platlet rich fibrin
- control group (Placebo Comparator)
  Interventions: Procedure: one side in control group

INTERVENTIONS:
Procedure: autologous platlet rich fibrin — one dose immediate after surgery
  Other Names: prf
  Arms: prf group.peridontal problem
Procedure: one side in control group — control group insert any things after surgery
  Arms: control group

SUMMARY:
The purpose of this study is to determine the influence of platelet rich fibrin to reduction of periodontal problems after surgical removal of third molar.

DETAILED DESCRIPTION:
After extraction or surgical removal of third molar, a deep bony pocket created behind the second molar specially in the mandible. For reduction of this problem, investigators, needed to acceleration tissue healing. For this purpose, investigators used platelet rich fibrin (autologous) and followed patient for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* have 2 impacted third molars

Exclusion Criteria:

* periodontal disease
* history of periodontal surgery

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Measurement of periodontal pocket depth at mid buccal, disto buccal and distolingual of mandibular second molar | 4 months